CLINICAL TRIAL: NCT04713800
Title: Randomized Controlled Clinical Trial of Two-unit Cantilever Implant Prostheses Made of Monolithic Zirconia on Titanium Base Abutments or Porcelain-fused to Metal on Gold Abutments
Brief Title: Two-unit Cantilever Implant Prostheses Made of Monolithic Zirconia or PFM
Acronym: Cantilever
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Collaborators: ITI Foundation (Industry)
Responsible Party: Principal Investigator, João Pitta, Principal Investigator, Research and Teaching Fellow, University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cantilver study
Record Dates: First submitted 2021-01-12; First posted 2021-01-19 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Jaw, Edentulous, Partially; Missing Teeth
Keywords: Dental Implants; Cantilever; Titanium base; Dental abutment; Fixed dental prosthesis; Monolithic zirconia; Porcelain fused to metal
MeSH Terms: conditions — Jaw, Edentulous, Partially; Anodontia | interventions — Crowns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ZR-TiB (Experimental): Monolithic zirconia screw retained implant-supported cantilever reconstruction supported by titanium base abutments, in a full digital workflow (ZR)
  Interventions: Device: Monolithic zirconia screw retained implant-supported cantilever reconstruction supported by titanium base abutments, in a full digital workflow (ZR-TiB)
- PFM-GA (Active Comparator): Porcelain fused-to metal screw retained implant-supported cantilever reconstruction supported by a gold-abutment, in a conventional workflow (PFM)
  Interventions: Device: porcelain fused-to metal screw retained implant-supported cantilever reconstruction supported by a gold-abutment, in a conventional workflow (PFM-GA)

INTERVENTIONS:
Device: Monolithic zirconia screw retained implant-supported cantilever reconstruction supported by titanium base abutments, in a full digital workflow (ZR-TiB) — In group ZR-TiB the implant impressions will be taken using an intra-oral scanner and the respective scanbody. The restorations will be manufactured by means of CAD/CAM procedures using monolithic zirconia. For sufficient aesthetics, the zirconia restorations can be manually veneered with veneering ceramic only at the buccal surface, while the occlusal surface will remain monolithic and will be high-gloss polished. The zirconia restorations will be extra-orally cemented onto titanium base abutments (Straumann® Variobase® for crown, Straumann AG), correctly polished and delivered to the patient, by screw-retention onto the implant.
  Other Names: Straumann® Variobase® for crown
  Arms: ZR-TiB
Device: porcelain fused-to metal screw retained implant-supported cantilever reconstruction supported by a gold-abutment, in a conventional workflow (PFM-GA) — In group PFM-GA implant impression will be taken using a polyvinyl siloxane or polyether impression material in a conventional manner with the use of stock trays and corresponding impression copings. The framework will be manufactured by the lost wax-technique using a gold-abutment (Straumann® Gold abutment for crown, Straumann AG) and a gold-alloy. All metal frameworks will be manually veneered with veneering ceramic, polished and glazed, and delivered to the patient, by screw-retention onto the implant.
  Other Names: Straumann® Gold abutment for crown
  Arms: PFM-GA

SUMMARY:
The aim of is to compare the survival rate and technical outcomes of cantilever implant-supported fixed denture prosthetics (cFDPs) made either out of monolithic zirconia bonded to a titanium base in a digital workflow, or porcelain fused-to metal using a gold abutment in a conventional workflow. In addition, biological outcomes, wear patterns, PROMs and time efficiency will be recorded. The null hypothesis is: the reconstruction type does not influence the survival rate and technical outcomes of 2-unit implant-supported cFDP.

ELIGIBILITY:
Inclusion Criteria:

* Minimal age of 22 years old.
* No general medical condition which represents a contraindication to implant treatment
* Good oral hygiene (PII ≤ 20%), and healthy periodontal tissues (BOP≤ 20%)
* Two adjacent-teeth gap in posterior maxilla or mandible arch (first premolar, second premolar, first molar, second molar) with an osseointegrated regular or wide-diameter bone-level implant in a prosthetically correct position to allow occlusal screw-retention. Free-end edentulous gaps can also be included
* Presence of antagonist occlusal units

Exclusion Criteria:

* Severe bruxism or clenching habits
* Patients with inadequate oral hygiene or persistent intraoral infection
* Women who are pregnant or breast feeding at the day of inclusion
* Smokers exceeding 15 cigarettes / day, or equivalent; patients chewing tobacco
* Unable or unwilling to cooperate for the trial period
* Estimated cantilever crown mesial-distal length > 10 mm
* Estimated implant crown height (from implant platform to occlusal contact points) > 15 mm

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Technical complication rate | 5 years
  assessed by USPHS-criteria

SECONDARY OUTCOMES:
Survival rate | 1, 3, 5 years
Biological parameters | 1, 3, 5 years
  assessed by clinical examination by measuring with a periodontal probe: bleeding on probing (yes/no per site), pocket probing depth (mm), width of keratinized mucosa (mm), assessed by evaluation of standardized x-rays: marginal bone level changes (mm)
Wear rate of restoration and antagonist | 1, 3, 5 years
  assessed by a volumetric analysis software
Patient Reported Outcomes Measures (PROMs) | 1, 3, 5 years
  assessed through questionnaires: Oral Health Impact Profile (OHIP-14) to evaluate oral health-related quality of life [0-4 for each of the 14 questions, where 4 represents the worst outcome]; Visual Analogue Scales (VAS) to evaluate patient experience with the impression procedure [0-10, where 10 represents the best outcome]
Cost-efficiency | single-point measure at baseline
  assessed by measuring time and counting costs of materials between the two workflows procedures (digital vs. analogue)
Accuracy of fabrication | single-point measure at baseline
  measured in terms of occlusal adjustment needed between the two fabrication procedures (digital vs. analogue workflow)
Operator Reported Outcomes Measures | single-point measure at baseline
  assessed through Visual Analogue Scales (VAS) to evaluate operator experience with the impression procedure and with the adjustment of the restoration [0-10, where 10 represents the best outcome]

CONTACTS AND LOCATIONS:
Overall Officials: João Pitta, Dr, Principal Investigator — University of Geneva; Irena Sailer, Prof, Study Chair — University of Geneva
Locations (1):
- University of Geneva, Geneva, Switzerland